CLINICAL TRIAL: NCT01168999
Title: The Mechanisms of Manual Therapy in the Treatment of Low Back Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 345-2009
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Low Back Pain
Keywords: low back pain; spinal manipulation; manual therapy; placebo
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- spinal manipulation (Active Comparator): a spinal manipulation known to be effective in the treatment of low back pain for some individuals
  Interventions: Other: spinal manipulation
- sham spinal manipulation (Placebo Comparator): a sham spinal manipulation intended to mimic the studied spinal manipulation
  Interventions: Other: sham spinal manipulation
- natural history (No Intervention): No intervention is provided to participants in this arm of the study
- Enhanced sham spinal manipulation (Placebo Comparator): a sham spinal manipulation intended to mimic the studied spinal manipulation and provided with the instructions, "The manual therapy technique you will receive has been shown to significantly reduce low back pain in some people"
  Interventions: Other: Enhanced sham spinal manipulation

INTERVENTIONS:
Other: spinal manipulation — Spinal manipulation commonly used in the treatment of low back pain and known to be effective for some individuals experiencing low back pain
  Arms: spinal manipulation
Other: sham spinal manipulation — Sham spinal manipulation intended to mimic the studied spinal manipulation
  Arms: sham spinal manipulation
Other: Enhanced sham spinal manipulation — Sham spinal manipulation intended to mimic the studied spinal manipulation and provided with the instructions, "The manual therapy technique you will receive has been shown to significantly reduce low back pain in some people"
  Arms: Enhanced sham spinal manipulation

SUMMARY:
The purpose of this study is to determine whether a novel placebo for comparison to spinal manipulation is believable and creates similar expectation for treatment effectiveness as the studied spinal manipulation technique. Additionally, we wish to compare outcomes related to low back pain, function, and pain sensitivity between people receiving the placebo, spinal manipulation, and no therapy.

ELIGIBILITY:
Inclusion Criteria:

* currently experiencing low back pain which does not extend below the knees
* rate the low back pain as a minimum of 4/10 at worst over the past 24 hours
* appropriate for conservative management of low back pain
* english speaking

Exclusion Criteria:

* surgery to the low back over the past 6 months
* systemic disease known to effect sensation
* other chronic pain condition unrelated to low back pain
* fracture as a cause of low back pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Bialosky, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Bialosky JE, George SZ, Horn ME, Price DD, Staud R, Robinson ME. Spinal manipulative therapy-specific changes in pain sensitivity in individuals with low back pain (NCT01168999). J Pain. 2014 Feb;15(2):136-48. doi: 10.1016/j.jpain.2013.10.005. Epub 2013 Oct 27. PMID 24361109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was undertaken in a lab on the University of Florida. Participants were recruited through written and electronic advertisement approved by the University of Florida Institutional Review Board. The first participant was enrolled in the study in November of 2009 and the final participant completed the study in January of 2013.
Groups:
- Spinal Manipulative Therapy: Received a spinal manipulative therapy commonly provided to individuals with low back pain for 6 sessions over 2 weeks
- Sham Spinal Manipulative Therapy: Received a sham spinal manipulative therapy for 6 sessions over 2 weeks.
- Enhanced Sham Spinal Manipulative Therapy: Received the sham spinal manipulative therapy with the instructional set The manual therapy technique you will receive has been shown to significantly reduce low back pain in some people for 6 sessions over 2 weeks.
- Natural History: These participants sat quietly for 5 minutes during the initial and final testing sessions.
Period: Overall Study
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Started | 28 | 27 | 27 | 28
Completed | 26 | 26 | 27 | 28
Not Completed | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History | Total
Number analyzed (Participants) | 28 | 27 | 27 | 28 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 27 | 28 | 110
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.07 (10.98) | 33.22 (13.29) | 31.56 (11.85) | 29.85 (12.09) | 31.68 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 20 | 19 | 77
  Male | 7 | 10 | 7 | 9 | 33
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 27 | 28 | 110

OUTCOME MEASURES:

1. Primary Outcome: Believability of Placebo
Description: Assess whether or not participants receiving the placebo are blinded to the fact they are receiving the placebo as indicated by the percentage of participants in each arm of the study believing they received SMT
Time Frame: baseline
Measure: Number; unit: percentage of participants
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Number analyzed (Participants) | 28 | 27 | 27 | 0
percentage of participants | 67 | 37 | 78 |
Statistical Analysis 1: Comparison: Spinal Manipulative Therapy vs Sham Spinal Manipulative Therapy vs Enhanced Sham Spinal Manipulative Therapy; Test type: Superiority or Other; p < 0.01, Chi-squared

2. Primary Outcome: Expectation for Treatment Effectiveness
Description: how helpful participants expect the assigned intervention will be in decreasing their low back pain
Time Frame: baseline
Measure: Number; unit: percent expecting less pain
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Number analyzed (Participants) | 28 | 27 | 27 | 28
percent expecting less pain | 54 | 26 | 59 | 11
Statistical Analysis 1: Comparison: Spinal Manipulative Therapy vs Sham Spinal Manipulative Therapy vs Enhanced Sham Spinal Manipulative Therapy vs Natural History; Test type: Superiority or Other; p = 0.01, Chi-squared

3. Primary Outcome: Change From Baseline at 2 Weeks in Clinical Pain as Measured by a Numeric Rating Scale
Description: A 101 point numeric rating scale with 0= no pain at all to 100= worst pain imaginable of low back pain
Time Frame: Change from Baseline at 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Number analyzed (Participants) | 26 | 26 | 27 | 28
units on a scale | 11.23 (14.01) | 14.03 (17.88) | 9.44 (25.90) | 8.20 (12.64)
Statistical Analysis 1: Comparison: Spinal Manipulative Therapy vs Sham Spinal Manipulative Therapy vs Enhanced Sham Spinal Manipulative Therapy vs Natural History; Test type: Superiority or Other; p > 0.05, Repeated Measure ANOVA

4. Primary Outcome: Change From Baseline at 2 Weeks in Disability as Measured by the Oswestry Disability Index
Description: The Oswestry Disability Index is a 10 item questionnaire measuring low back pain related disability. Individual item scores range from 0 to 5. Scores on all items are summed and multiplied by 2 to provide a percentage ranging between 0 to 100 with higher scores indicating greater low back pain related disability.
Time Frame: Change from Baseline at 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Number analyzed (Participants) | 26 | 26 | 27 | 28
units on a scale | 4.46 (8.28) | 2.08 (7.36) | 2.69 (8.33) | 2.54 (8.47)
Statistical Analysis 1: Comparison: Spinal Manipulative Therapy vs Sham Spinal Manipulative Therapy vs Enhanced Sham Spinal Manipulative Therapy vs Natural History; Test type: Superiority or Other; p > 0.05, Repeated Measure ANOVA

5. Primary Outcome: Change in Pain Sensitivity From Baseline to Immediately Following the Assigned Intervention as Measured by a Visual Analog Scale
Description: Participants received a standard thermal stimulus to the bottom of their foot prior to and immediately following their assigned intervention. Participants rated their pain in response to this thermal stimulus using a 101 mm visual analog scale with 0 mm indicating "no pain at all" and 100 mm indicating "the worst pain imaginable".
Time Frame: baseline and immediately following their assigned intervention during the initial session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Number analyzed (Participants) | 28 | 27 | 27 | 28
units on a scale | 8.14 (20.48) | -3.04 (12.92) | 1.22 (16.03) | -2.93 (17.84)
Statistical Analysis 1: Comparison: Spinal Manipulative Therapy vs Sham Spinal Manipulative Therapy vs Enhanced Sham Spinal Manipulative Therapy vs Natural History; Test type: Superiority or Other; p = 0.05, Repeated Measure ANOVA

6. Secondary Outcome: Change From Baseline at 2 Weeks in Low Back Flexion Range of Motion
Description: Low back flexion range of motion was measured in degrees using a gravity inclinometer
Time Frame: Change from Baseline at 2 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Number analyzed (Participants) | 26 | 26 | 27 | 28
degrees | 1.58 (8.65) | 2.67 (13.91) | -0.33 (9.55) | -0.54 (9.25)
Statistical Analysis 1: Comparison: Spinal Manipulative Therapy vs Sham Spinal Manipulative Therapy vs Enhanced Sham Spinal Manipulative Therapy vs Natural History; Test type: Superiority or Other; p > 0.05, Repeated Measure ANOVA

7. Secondary Outcome: Change From Baseline at 2 Weeks in Low Back Extension Range of Motion
Description: Low back extension range of motion was measured in degrees using a gravity inclinometer
Time Frame: Change from Baseline at 2 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Number analyzed (Participants) | 26 | 26 | 27 | 28
degrees | -1.50 (9.58) | -0.07 (11.26) | 1.26 (4.95) | -0.21 (7.82)

8. Secondary Outcome: Change From Baseline at 2 Weeks in Low Back Right Sidebending Range of Motion
Description: Low back right sidebending range of motion was measured in degrees using a gravity inclinometer
Time Frame: Change from Baseline at 2 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Number analyzed (Participants) | 26 | 26 | 27 | 28
degrees | 0.92 (8.68) | -0.19 (1.24) | 0.63 (7.53) | 0.50 (9.50)

9. Secondary Outcome: Change From Baseline at 2 Weeks in Low Back Left Sidebending Range of Motion
Description: Low back left sidebending range of motion was measured in degrees using a gravity inclinometer
Time Frame: Change from Baseline at 2 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Number analyzed (Participants) | 26 | 26 | 27 | 28
degrees | 2.15 (8.04) | -0.15 (6.37) | 1 (6.66) | -1.36 (6.41)

ADVERSE EVENTS:
Time Frame: The study was conducted from November of 2009 until January of 2013. The occurrence of adverse events was monitored during the length of the study.
Arm/Group | Spinal Manipulative Therapy | Sham Spinal Manipulative Therapy | Enhanced Sham Spinal Manipulative Therapy | Natural History
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes